CLINICAL TRIAL: NCT01348308
Title: Optimized Phase III Trial of Immuno-stimulation With Maraviroc, a CCR5 (Chemokine Receptor 5) Antagonist, Combined With Anti Retroviral Therapy in Advanced, Late Diagnosed HIV-1 Infected Patients With an AIDS-defining Event and/or CD4 (Cluster of Differentiation 4) Counts Below 200 Cells/mm³. ANRS 146 OPTIMAL
Brief Title: Immuno-stimulation With Maraviroc Combined to Antiretroviral Therapy in Advanced Late Diagnosed HIV-1 Infected Patients
Acronym: OPTIMAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2010-022293-14; ANRS 146 OPTIMAL
Record Dates: First submitted 2011-05-02; First posted 2011-05-05 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: HIV-1 Infection; AIDS
Keywords: Late diagnosed HIV-1 infected patients; AIDS-defining events; Immune restoration
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Maraviroc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Maraviroc (Active Comparator): Maraviroc 300, 600 or 1200mg per day
  Interventions: Drug: Maraviroc (Celsentri)
- Placebo (Placebo Comparator): Placebo 300, 600 or 1200mg per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Maraviroc (Celsentri) — Patients will take cART optimized regimen according to the recommended regimen as first line of treatment in most commonly used guidelines with Maraviroc at the following dose: 150 mg orally twice a day for patients receiving a Protease Inhibitor Ritonavir-boosted regimen (except Fosamprenavir), 300 mg orally twice a day for patients receiving a Fosamprenavir Ritonavir-boosted regimen or 600 mg orally twice a day for patients receiving Efavirenz-based regimen.
  Duration: 72 weeks.
  Arms: Maraviroc
Drug: Placebo — Patients will take cART optimized regimen according to the recommended regimen as first line of treatment in most commonly used guidelines with Placebo at the following dose: 150 mg orally twice a day for patients receiving a Protease Inhibitor Ritonavir-boosted regimen (except Fosamprenavir), 300 mg orally twice a day for patients receiving a Fosamprenavir Ritonavir-boosted regimen or 600 mg orally twice a day for patients receiving Efavirenz-based regimen.
  Duration: 72 weeks.
  Arms: Placebo

SUMMARY:
The objective of the OPTIMAL study is to demonstrate that the adjunction of Maraviroc to a combination of antiretroviral therapy in naive and late diagnosed HIV-1 infected patients counts may accelerate the kinetics of immune restoration and decrease the risk of disease progression and death.

It is a randomized, versus placebo, double-blind trial, conducted in France, Spain and Italy.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV-1 infection (ELISA and Western Blot tests positive)
* CD4+ T lymphocytes below or equal 200/mm³ or previous AIDS-defining-illness at diagnosis
* Patient naïve from any antiretroviral
* In women, use of a contraceptive method, and lack of actual pregnancy
* Patients with a coverage from social health
* After informed consent

Exclusion Criteria:

* Current pregnancy, lack of contraceptive method, breast-feeding
* Current active tuberculosis (either suspected, diagnosed)
* Ongoing malignancies except cutaneous Kaposi's sarcoma. Patients with a previous cancer considered as cured for at least 6 months could be included in the study
* Current or previous severe cardiac failure, chronic respiratory disease, renal or liver insufficiency; any life-threatening organ failure
* Cognitive impairment, psychiatric disorders, severe depressive affects, unadapted behavior
* Use of cytostatic drugs, immunosuppressive agents, steroids
* PMN (polymorphonuclear neutrophil) below 750/mm³, platelets below 50,000/mm³, haemoglobin below 10 g/dL; ASAT (aspartate aminotransferase), ALAT (alanine aminotransferase) or bilirubin over 2.5 ULN; lipase over 2 ULN (Upper limit of normal), serum creatinine over 1.5 ULN; proteinuria over 1g/L; INR (International Normalized Ratio) abnormal
* Current or previous, during the 3 last months, use of immunomodulatory agents (G-CSF (granulocyte colony stimulating factor), IL-2 (Interleukin-2), GM-CSF (Granulocyte Macrophage colony stimulating factor), interferons, pentoxifylline)
* Hypersensitivity to peanut and /or soy products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2011-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
To demonstrate the clinical benefit of the adjunction of Maraviroc to a combination of antiretroviral therapy defined as decrease of clinical events | From Week 0 to Week 72
  The clinical benefit is the reduction of occurence of a composite outcome consisting of:
  * New AID-defining event (1993 CDC(Centers for Disease Control) expanded surveillance definition)
  * Non B or C events (Aspergillosis, Bartonellosis, Chagas disease, Leishmaniasis, Lymphoma, Microsporidiosis chronic intestinal, Nocardiosis, Penicillium marneffei extrapulmonary, Pneumocystis jiroveci extrapulmonary, Rhodococcus equi disease, Severe bacterial infections)
  * Serious non-AIDS events (Cardiovascular disease, Chronic end stage renal disease, Liver failure, Non-AIDS defining cancers, IRIS)
  * All cause of mortality

SECONDARY OUTCOMES:
Safety evaluation and Clinical, Immunological and pharmacological evaluation | From Week 0 to Week 72
  The secondary end points:
  * Clinical events (to compare Maraviroc and placebo arm for each component of the primary composite endpoint and other major outcomes)
  * Immunological evaluation (T cells phenotypic analysis; seric markers of immune activation)
  * Virological evaluation (plasma HIV viral load analysis; viral tropism testing,)
  * Pharmacokinetic evaluation (plasma concentration of Maraviroc and relationship with virological response)
  * Clinical and biological safety of the strategy (Adverse events >= grade 2 on ANRS scale of adverse event)
  * Cost-effectiveness analysis

CONTACTS AND LOCATIONS:
Overall Officials: Yves Levy, MD, PhD, Study Chair — APHP, Hopital Henri Mondor, Creteil, France; Jean-Daniel Lelievre, MD, PhD, Principal Investigator — APHP, Hopital Henri Mondor, Creteil, France; Dominique Costagliola, PhD, Study Director — INSERM U943 and Univerité Pierre et Marie Curie
Locations (1):
- Hôpital Henri Mondor, Créteil, France

REFERENCES:
- [Derived] Levy Y, Lelievre JD, Assoumou L, Aznar E, Pulido F, Tambussi G, Crespo M, Meybeck A, Molina JM, Delaugerre C, Izopet J, Peytavin G, Cardon F, Diallo A, Lancar R, Beniguel L, Costagliola D. Addition of Maraviroc Versus Placebo to Standard Antiretroviral Therapy for Initial Treatment of Advanced HIV Infection: A Randomized Trial. Ann Intern Med. 2020 Mar 3;172(5):297-305. doi: 10.7326/M19-2133. Epub 2020 Feb 11. PMID 32040959
- See also: Related Info — http://www.anrs.fr/